CLINICAL TRIAL: NCT06708494
Title: Establishing Video Decision Aids for Geriatric Patients With Frailty to Promote Advance Care Planning: Comprehensibility, Usability, Feasibility
Brief Title: Establishing Video Decision Aids for Geriatric Patients With Frailty to Promote Advance Care Planning
Status: Enrolling by invitation | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202403006RIFC
Record Dates: First submitted 2024-11-20; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-03

CONDITIONS: Frailty
Keywords: Frailty; Advance Care Planning; Video Decision Aids
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: video decision aids — The video includes an introduction to geriatric frailty (3 minutes) and ACP (5 minutes). ACP includes three levels of medical care: life-prolonging care, limited care, and comfort care.

SUMMARY:
The goal of this observational study aimed to develop and assess a video decision aid for advance care planning in geriatric patients with frailty. The main question it aims to answer is:

The video decision aid comprehensibility, usability, feasibility? The video includes an introduction to geriatric frailty (3 minutes) and advance care planning (5 minutes). Advance care planning includes three levels of medical care: life-prolonging care, limited care, and comfort care.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1 - Patients

  1. Aged 65 or older.
  2. Have not completed an advance directive (AD) document.
  3. Able to communicate in Mandarin or Taiwanese.
  4. Have adequate vision and hearing to watch a video in Mandarin or Taiwanese on a tablet.
  5. Willing to participate in the study after explanation.
* Phase 1 - Family Members

  1. Aged 18 or older.
  2. Have not completed an advance directive (AD) document.
  3. Able to communicate in Mandarin or Taiwanese.
  4. Have adequate vision and hearing to watch a video in Mandarin or Taiwanese on a tablet.
  5. Willing to participate in the study after explanation.
* Phase 1 - Healthcare Providers

  1. Have not completed an advance directive (AD) document.
  2. Able to communicate in Mandarin or Taiwanese.
  3. Willing to participate in the study after explanation.
* Phase 2 - Patients

  1. Aged 65 or older.
  2. Have participated in shared decision-making (SDM) using decision aid tools.
  3. Have experience in advance care planning (ACP) consultation or have completed related written advance directive documents.
  4. Able to communicate in Mandarin or Taiwanese.
  5. Have adequate vision and hearing to watch a video in Mandarin or Taiwanese on a tablet.
  6. Willing to participate in the study after explanation.
* Phase 2 - Healthcare Providers

  1. Have professional knowledge and practical experience in advance care planning (ACP).
  2. Have experience caring for frail elderly populations.
  3. Able to communicate in Mandarin or Taiwanese.
  4. Willing to participate in the study after explanation.

Exclusion Criteria:

1.Cognitive impairment, unable to communicate clearly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: National Taiwan University Hospital inpatient wards or the Department of Family Medicine's Geriatric Frailty Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
comprehensibility | Watching a 10-minute video and completing questionnaire takes approximately 5-10 minutes.
  Comprehensibility was measured using a knowledge questionnaire and the Patient Education Materials Assessment Tool for Audiovisual Materials (PEMAT-A/V).The knowledge questionnaire consists of 7 questions, each with 10 correct answer choices, scored at 10 points per correct choice, for a total of 100 points. Higher scores indicate greater accuracy in knowledge and better comprehension. The PEMAT-A/V evaluates comprehension through 13 items and feasibility through 4 items. Responses are scored as Agree = 1 point, Disagree = 0 points, and Not Applicable (N/A) excluded from the total score calculation. The final score is calculated as Total Points/Total Possible Points x 100. Higher scores indicate that the material is easier to comprehend or more feasibility.
  Measurement timing: elder patients and their family members will complete the knowledge questionnaire before viewing the video. They will also complete the PEMAT A/V within one hour after viewing the materials.
usability | Watching a 10-minute video and completing questionnaire takes approximately 5-10 minute
  Usability was evaluated through a feedback questionnaire. The feedback questionnaire consists of 6 items. Except for the final open-ended question, the remaining items are scored using a 4-point Likert scale (0-3). Lower scores indicate higher usability.
  Measurement timing: elder patients and their family members will complete the feedback questionnaire within one hour after viewing the materials.
feasibility | Watching a 10-minute video and completing questionnaire takes approximately 5-10 minute
  Feasibility were evaluated through the PEMAT-A/V. The PEMAT-A/V evaluates comprehension through 13 items and feasibility through 4 items. Responses are scored as Agree = 1 point, Disagree = 0 points, and Not Applicable (N/A) excluded from the total score calculation. The final score is calculated as Total Points/Total Possible Points x 100. Higher scores indicate that the material is easier to comprehend or more feasibility.
  Measurement timing: elder patients and Healthcare professionals (Have experience in advance care planning) will complete the PEMAT A/V within one hour after viewing the materials.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No